CLINICAL TRIAL: NCT02060383
Title: A Multi-center, Randomized, Open-label, Phase IV Study to Investigate the Management of Pasireotide-induced Hyperglycemia With Incretin Based Therapy or Insulin in Adult Patients With Cushing's Disease or Acromegaly
Brief Title: Study of Management of Pasireotide-induced Hyperglycemia in Adult Patients With Cushing's Disease or Acromegaly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CSOM230B2219; 2012-002916-16 (EudraCT Number)
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Cushing's Disease; Acromegaly
Keywords: Cushing's disease; acromegaly; pasireotide; hyperglycemia
MeSH Terms: conditions — Pituitary ACTH Hypersecretion; Acromegaly; Hyperglycemia | interventions — pasireotide; Sitagliptin Phosphate; Liraglutide; Insulin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Incretin based therapy (randomized group) (Experimental): Participants randomized to the incretin based arm started with sitagliptin once daily. If sitagliptin did not control the participant's hyperglycemia, sitagliptin was stopped and participants switched to liraglutide once daily. If despite treatment with liraglutide, hyperglycemia was not controlled then the participant was eligible for rescue therapy with addition of insulin.
  Interventions: Drug: Pasireotide s.c.; Drug: Sitagliptin; Drug: Liraglutide; Drug: Insulin; Drug: Pasireotide LAR; Drug: Metformin
- Insulin (randomized group) (Experimental): Participants randomized to the insulin arm started with once daily dose of basal insulin. The dose was up or down titrated at the discretion of the investigator. If blood glucose levels remained uncontrolled on basal insulin, participant switched to basal insulin plus prandial insulin.
  Interventions: Drug: Pasireotide s.c.; Drug: Insulin; Drug: Pasireotide LAR; Drug: Metformin
- Non-Randomized Arm (Other): This arm represents the non-randomized participants: Cushing's Disease (CD) or Acromegaly participants, who received pasireotide s.c. or LAR (long-acting release) respectively, but who were not randomized to the Incretin or Insulin arms.
  For the purpose of analysis, this non-randomized arm is further split into 3 groups:
  * Baseline insulin group (BL insulin) includes participants who were receiving insulin at study entry
  * Oral antidiabetic drugs (OAD) group includes participants who developed hyperglycemia that was controlled by metformin and/or other background anti-diabetic treatment
  * No OAD group includes participants who did not receive any anti-diabetic medication during the core phase of the trial
  Interventions: Drug: Pasireotide s.c.; Drug: Insulin; Drug: Pasireotide LAR; Drug: Metformin

INTERVENTIONS:
Drug: Pasireotide s.c. — Administered to Cushing's disease participants.
  Other Names: SOM230
Drug: Sitagliptin — Taken for approximately 16 weeks during the core study phase or until the drug was found not to be effective
  Arms: Incretin based therapy (randomized group)
Drug: Liraglutide — Participant switched to liraglutide if sitagliptin was found not to be effective.
  Arms: Incretin based therapy (randomized group)
Drug: Insulin — Participant took insulin for 16 weeks. Insulin was also administered as rescue therapy in the incretin-based therapy arm if required.
  Insulin was administered to the BL-insulin group at the discretion of the Principal Investigator.
  Note: OAD and No OAD groups within the non-randomized arm did not take Insulin.
Drug: Pasireotide LAR — Administered to Acromegaly participants.
  Other Names: SOM230
Drug: Metformin — If previously normo-glycemic participants experienced increase in their fasting blood glucose and meeting the criteria for diabetes while on pasireotide, they started anti-diabetic treatment using metformin. If they continued to experience increase in their fasting blood glucose within the first 16 weeks, they were randomized in a 1:1 ratio to receive treatment with incretin based therapy or insulin for approximately 16 weeks. Metformin treatment was not required for the BL Insulin and OAD groups, within the non-randomized arm, but may have been prescribed at the discretion of the investigator.
  Note: No OAD group within the non-randomized arm did not take metformin.

SUMMARY:
The study was designed to investigate the optimal management of hyperglycemia developed during pasireotide treatment in participants with Cushing's disease or Acromegaly, which was not manageable with metformin.

This was a Phase IV, multi-center, randomized, open-label study. Eligible patients started pasireotide subcutaneously (s.c.) for Cushing's disease and pasireotide LAR (long-acting release) for Acromegaly.

Participants being treated with pasireotide s.c or LAR at screening were eligible as long as they met protocol criteria during the screening period. If previously normo-glycemic participants experienced an increase in their fasting blood glucose and met the criteria for diabetes while on pasireotide, they started anti-diabetic treatment using metformin. If they continued to have elevated blood glucose above target on metformin within the first 16 weeks, they were randomized in a 1:1 ratio to receive treatment with incretin based therapy or insulin for approximately 16 weeks.

Participants who continued to receive clinical benefit after completing the Core Phase could enter an optional Extension Phase if pasireotide was not commercially available in their country or a local access program was not available to provide drug. Patients continued in the Extension Phase until the last participant randomized in the Core Phase completed 16 weeks of treatment post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than or equal to 18 years old
* Confirmed diagnosis of Cushing's disease or acromegaly

Exclusion Criteria:

* Patients who require surgical intervention
* Patients receiving DPP-4 inhibitors or GLP-1 receptor agonists within 4 weeks prior to study entry
* HbA1c > 10 % at screening
* Known hypersensitivity to somatostatin analogues Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (42):
- United States (15):
  - Diabetes and Endocrine Associates La Mesa Location, Multiple Locations, California
  - LA Biomedical Research at Harbor UCLA Medical Center SC - SOM230B2219, Torrance, California
  - Coastal Metabolic Research Centre SC, Ventura, California
  - East Coast Institute for Research East Coast Inst. for Res(ECIR), Jacksonville, Florida
  - Washington University SC - SOM230B2411, St Louis, Missouri
  - Great Falls Clinic, Great Falls, Montana
  - Robert Wood Johnson Medical School - Rutgers SC, New Brunswick, New Jersey
  - The Mount Sinai Hospital SC, New York, New York
  - Columbia University Medical Center New York Presbyterian Neuroendocrine Unit, New York, New York
  - Lenox Hill Hospital/Manhattan Eye, Ear and Throat Hospital SC, New York, New York
  - Allegheny Endocrinology Associates SC, Pittsburgh, Pennsylvania
  - Vanderbilt Clinical Trials Center SOM230B2219, Nashville, Tennessee
  - Baylor College of Medicine Ben Taub General Hosp., Houston, Texas
  - Virginia Endocrinology Research SC-2, Chesapeake, Virginia
  - Swedish Medical Center Dept.ofSeattle Neuroscience(2), Seattle, Washington
- Belgium (2):
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Wilrijk
- Brazil (4):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Joinville, Santa Catarina
  - Novartis Investigative Site, São Paulo, São Paulo
- China (3):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Chengdu, Sichuan
- Denmark (4):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Odense C
- Germany (3):
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Oldenburg
- India (2):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Vellore, Tamil Nadu
- Novartis Investigative Site, San Isidro, Lima region, Peru
- Poland (2):
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, Saint Petersburg, Russia
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Songkhla
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Altunizade
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Antalya

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Samson SL, Gu F, Feldt-Rasmussen U, Zhang S, Yu Y, Witek P, Kalra P, Pedroncelli AM, Pultar P, Jabbour N, Paul M, Bolanowski M. Managing pasireotide-associated hyperglycemia: a randomized, open-label, Phase IV study. Pituitary. 2021 Dec;24(6):887-903. doi: 10.1007/s11102-021-01161-4. Epub 2021 Jul 18. PMID 34275099
- [Derived] Silverstein JM. Hyperglycemia induced by pasireotide in patients with Cushing's disease or acromegaly. Pituitary. 2016 Oct;19(5):536-43. doi: 10.1007/s11102-016-0734-1. PMID 27405306

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 68 randomized evaluable participants with at least 8 weeks of randomized treatment without any rescue anti-diabetic medication was required. Approximately 79 participants were planned to be randomized.
Pre-assignment Details: 249 participants were included in study & treated with pasireotide s.c. (59 with Cushing's disease) or pasireotide LAR (190 with acromegaly). Following pre-randomization period (up to 16 weeks), 81 participants were randomized to either incretin-based therapy or insulin (72 evaluable for the primary analysis) & 168 not qualified for randomization.
Groups:
- Baseline Insulin (BL) (Non-randomized Group): This group included participants who were receiving insulin at study entry.
- Oral Antidiabetic Drugs (OAD) (Non-randomized Group): This group included participants who developed hyperglycemia that was controlled by metformin and/or other background anti-diabetic treatment. Patients in this group did not require additional treatment with either incretin or insulin.
- No OAD (Non-randomized Group): This group included participants who did not receive any anti-diabetic medication during the Core Phase of the study as they did not develop hyperglycemia.
Period: Core Phase
Arm/Group | Incretin Based Therapy (Randomized Group) | Insulin (Randomized Group) | Baseline Insulin (BL) (Non-randomized Group) | Oral Antidiabetic Drugs (OAD) (Non-randomized Group) | No OAD (Non-randomized Group)
Started (Entered Core Phase of Study) | 38 | 43 | 19 | 46 | 103
Completed Core/Entered Extension | 17 | 17 | 10 | 21 | 53
Completed Core/Did Not Enter Extension | 18 | 20 | 9 | 18 | 42
Completed | 35 | 37 | 19 | 39 | 95
Not Completed | 3 | 6 | 0 | 7 | 8
Not completed — Unsatisfactory therapeutic effect | 1 | 5 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 2 | 6
Not completed — Administrative problems | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4 | 2
Period: Extension Phase
Arm/Group | Incretin Based Therapy (Randomized Group) | Insulin (Randomized Group) | Baseline Insulin (BL) (Non-randomized Group) | Oral Antidiabetic Drugs (OAD) (Non-randomized Group) | No OAD (Non-randomized Group)
Started (Entered the Extension phase from the Core phase) | 17 | 17 | 10 | 21 | 53
Completed (Completed the Extension phase) | 14 | 14 | 7 | 19 | 46
Not Completed | 3 | 3 | 3 | 2 | 7
Not completed — Unsatisfactory therapeutic effect | 1 | 1 | 0 | 2 | 2
Not completed — Adverse Event | 1 | 1 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 2
Not completed — Administrative problems | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants who received at least one dose of pasireotide.
Groups:
- Total: Total of all reporting groups
Arm/Group | Incretin Based Therapy (Randomized Group) | Insulin (Randomized Group) | Baseline Insulin (BL) (Non-randomized Group) | Oral Antidiabetic Drugs (OAD) (Non-randomized Group) | No OAD (Non-randomized Group) | Total
Number analyzed (Participants) | 38 | 43 | 19 | 46 | 103 | 249
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.6 (11.76) | 46.4 (12.90) | 46.7 (12.54) | 40.2 (13.80) | 37.8 (11.17) | 42.4 (13.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 10 | 31 | 47 | 137
  Male | 16 | 16 | 9 | 15 | 56 | 112
Race/Ethnicity, Customized [Number; unit: Participants]
  Other | 22 | 24 | 11 | 25 | 43 | 125
  Chinese | 5 | 9 | 1 | 13 | 33 | 61
  Hispanic/Latino | 7 | 2 | 5 | 6 | 19 | 39
  Indian (Indian subcontinent) | 4 | 8 | 2 | 2 | 7 | 23
  Japanese | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Randomization to Approximately 16 Weeks
Description: Absolute change in HbA1c from randomization to end of core phase (16 weeks) in incretin based therapy arm and insulin arm, and mean difference of change in HbA1c between the two treatment groups based on an ANOVA model using treatment (Incretin, Insulin) and the two randomization stratification factors (Disease: Cushing's disease vs Acromegaly; Baseline glycemic status: HbA1c <7% vs HbA1c ≥ 7%) as fixed effects. For Participants who discontinued the study or required rescue treatment before the time of assessing the primary endpoint, the last HbA1c assessment collected 8 weeks (56 days) after randomization (and prior to or on the date of start of rescue treatment) was carried forward. If the participant discontinued the study or used rescue treatment within 8 weeks after randomization, it was considered missing.
Time Frame: Randomization, 16 weeks
Population: Randomized Analysis Set (RAS): all patients who received at least one dose of pasireotide and were assigned to either incretin based therapy or insulin by randomization.
  If the patient discontinued the study or used rescue treatment within 8 weeks after randomization, it was considered missing.
Measure: Mean (95% Confidence Interval); unit: Hba1c percentage
Arm/Group | Incretin Based Therapy (Randomized Group) | Insulin (Randomized Group)
Number analyzed (Participants) | 31 | 41
Hba1c percentage
  All Patients | -0.12 [-0.36 to 0.13] | 0.26 [-0.01 to 0.53]
  Cushing's Disease: number analyzed (Participants) | 7 | 11
  Cushing's Disease | 0.33 [-0.41 to 1.07] | 0.45 [-0.20 to 1.09]
  Acromegaly: number analyzed (Participants) | 24 | 30
  Acromegaly | -0.25 [-0.49 to -0.00] | 0.19 [-0.12 to 0.49]
Statistical Analysis 1: Comparison: Incretin Based Therapy (Randomized Group) vs Insulin (Randomized Group); All Patients; Test type: Other — There was no formal hypothesis testing planned in this study; Mean Difference (Net) = -0.28, 95% CI 2-sided [-0.63 to 0.08], Standard Error of Mean 0.18 — Difference of adjusted mean change in HbA1c between the two arms based on an ANOVA model with treatment (Incretin, Insulin) and randomization stratification factors (Cushing's vs. Acromegaly; baseline HbA1c <7% vs ≥7%) as fixed effects
Statistical Analysis 2: Comparison: Incretin Based Therapy (Randomized Group) vs Insulin (Randomized Group); Cushing's Disease; Test type: Other — There was no formal hypothesis testing planned in this study; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.96 to 0.95], Standard Error of Mean 0.45 — Difference of adjusted mean change in HbA1c between the two arms based on an ANOVA model with treatment (Incretin, Insulin) and randomization stratification factors (baseline HbA1c <7% vs ≥7%) as fixed effects
Statistical Analysis 3: Comparison: Incretin Based Therapy (Randomized Group) vs Insulin (Randomized Group); Acromegaly; Test type: Other — There was no formal hypothesis testing planned in this study; Mean Difference (Net) = -0.36, 95% CI 2-sided [-0.74 to 0.02], Standard Error of Mean 0.19 — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Change in HbA1c From Randomization (R) Over Time Per Randomized Arm
Description: Absolute change in HbA1c overtime from randomization (i.e. start of randomized antidiabetic treatment) to end of core phase per randomized arm
Time Frame: Randomization (R), Week (W) 4 post R, W 8 post R, W 16 post R, end of Core phase (up to week 16 post R)
Population: Randomized Analysis Set (RAS): all patients who received at least one dose of pasireotide and were assigned to either incretin based therapy or insulin by randomization.
Measure: Mean (Standard Deviation); unit: HbA1c percentage
Arm/Group | Incretin Based Therapy (Randomized Group) | Insulin (Randomized Group)
Number analyzed (Participants) | 38 | 43
HbA1c percentage
  Randomization | 7.1 (1.00) | 7.1 (0.75)
  Change at RW4 D29: number analyzed (Participants) | 37 | 43
  Change at RW4 D29 | 0.5 (0.73) | 0.5 (0.60)
  Change at RW8 D57: number analyzed (Participants) | 37 | 43
  Change at RW8 D57 | 0.3 (0.98) | 0.5 (0.86)
  Change at RW12 D85: number analyzed (Participants) | 37 | 40
  Change at RW12 D85 | 0.2 (1.03) | 0.4 (0.85)
  Change at RW16 D113: number analyzed (Participants) | 35 | 37
  Change at RW16 D113 | 0.0 (0.93) | 0.3 (0.87)
  End of Core Phase: number analyzed (Participants) | 37 | 42
  End of Core Phase | 0.0 (0.92) | 0.3 (0.84)

3. Secondary Outcome: Change in FPG (Fasting Plasma Glucose) From Randomization Until End of Core Phase
Description: Absolute change in fasting glucose overtime from randomization (i.e. start of randomized antidiabetic treatment) to end of core phase per randomized arm
Time Frame: Randomization, R(randomization) Week 2, R-Week 4, R-Week 6, R-Week 8, R-Week 10, R-Week 12, R-Week 14, R-Week 16, end of Core phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Incretin Based Therapy (Randomized Group) | Insulin (Randomized Group)
Number analyzed (Participants) | 38 | 43
mg/dL
  Randomization | 172.2 (60.78) | 167.9 (40.77)
  Change at RW2 D15: number analyzed (Participants) | 36 | 42
  Change at RW2 D15 | 4.6 (51.01) | -31.1 (41.19)
  Change at RW4 D29 | -15.0 (47.95) | -28.3 (41.14)
  Change at RW6 D43: number analyzed (Participants) | 36 | 41
  Change at RW6 D43 | -17.7 (57.97) | -37.5 (52.39)
  Change at RW8 D57: number analyzed (Participants) | 36 | 42
  Change at RW8 D57 | -25.7 (53.32) | -38.3 (44.10)
  Change at RW10 D71: number analyzed (Participants) | 37 | 37
  Change at RW10 D71 | -28.8 (61.14) | -36.9 (50.82)
  Change at RW12 D85: number analyzed (Participants) | 37 | 40
  Change at RW12 D85 | -33.4 (50.17) | -41.1 (51.68)
  Change at RW14 D99: number analyzed (Participants) | 36 | 36
  Change at RW14 D99 | -35.1 (55.83) | -35.6 (47.43)
  Change at RW16 D113: number analyzed (Participants) | 35 | 34
  Change at RW16 D113 | -38.8 (53.69) | -33.4 (47.63)
  End of Core Phase: number analyzed (Participants) | 37 | 41
  End of Core Phase | -40.1 (56.35) | -36.0 (46.90)

4. Secondary Outcome: Percentage of Participants in the Incretin-based Arm Who Required Anti-diabetic Rescue Therapy With Insulin
Description: The percentage of participants who received anti-diabetic rescue therapy in incretin based therapy is summarized.
Time Frame: Randomization to up to 16 weeks
Population: Safety set - All participants randomized to the incretin-based therapy who received at least one dose of pasireotide and had at least one post-baseline safety assessment. Randomized participants within the safety set were analyzed according to the anti-diabetic study treatment first received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Incretin Based Therapy (Randomized Group)
Number analyzed (Participants) | 38
Percentage of participants | 31.6 [17.5 to 48.7]

5. Secondary Outcome: Absolute Change in HbA1c From Baseline to End of Core Phase
Description: Absolute change in HbA1c from baseline to end of core phase in the incretin based therapy arm and the insulin arm
Time Frame: Baseline, up to 32 weeks (end of Core phase)
Population: Full Analysis Set (FAS): Participants who received at least 1 dose of pasireotide. Randomized participants were analyzed according to the anti-diabetic treatment assigned to at randomization. Non-randomized participants were analyzed by the anti-diabetic treatment received during the core phase (insulin at baseline, oral antidiabetics (OAD), none).
Measure: Mean (Standard Deviation); unit: HbA1c percentage
Arm/Group | Incretin Based Therapy (Randomized Group) | Insulin (Randomized Group) | Baseline Insulin (BL) (Non-randomized Group) | Oral Antidiabetic Drugs (OAD) (Non-randomized Group) | No OAD (Non-randomized Group)
Number analyzed (Participants) | 38 | 43 | 19 | 46 | 103
HbA1c percentage
  Baseline: All Patients: number analyzed (Participants) | 38 | 43 | 19 | 46 | 102
  Baseline: All Patients | 6.3 (0.80) | 6.3 (0.63) | 7.7 (1.51) | 5.7 (0.41) | 5.4 (0.33)
  Change at EOP: All Patients: number analyzed (Participants) | 37 | 42 | 19 | 45 | 100
  Change at EOP: All Patients | 0.8 (0.97) | 1.1 (0.94) | 1.3 (1.40) | 0.8 (0.64) | 0.4 (0.32)
  Baseline: Cushing's: number analyzed (Participants) | 12 | 13 | 6 | 13 | 15
  Baseline: Cushing's | 6.6 (0.87) | 6.5 (0.58) | 6.9 (0.92) | 5.9 (0.49) | 5.5 (0.41)
  Change at EOP: Cushing's: number analyzed (Participants) | 12 | 13 | 6 | 13 | 14
  Change at EOP: Cushing's | 1.3 (1.19) | 1.7 (1.05) | 1.4 (1.58) | 0.9 (0.95) | 0.5 (0.51)
  Baseline: Acromegaly: number analyzed (Participants) | 26 | 30 | 13 | 33 | 87
  Baseline: Acromegaly | 6.1 (0.71) | 6.3 (0.65) | 8.0 (1.61) | 5.6 (0.36) | 5.4 (0.32)
  Change at EOP: Acromegaly: number analyzed (Participants) | 25 | 29 | 13 | 32 | 86
  Change at EOP: Acromegaly | 0.6 (0.78) | 0.8 (0.78) | 1.2 (1.37) | 0.7 (0.47) | 0.4 (0.28)

6. Secondary Outcome: Absolute Change in FPG From Baseline to End of Core Phase
Description: Absolute change in FPG from baseline to end of core phase in the incretin based therapy arm and the insulin arm.
Time Frame: Baseline, Up to 32 weeks (end of Core Phase)
Population: Full Analysis Set (FAS): All participants who received at least one dose of pasireotide. Randomized patients were analyzed according to the anti-diabetic treatment assigned to at randomization. Non-randomized patients were analyzed by the anti-diabetic treatment received during the core phase (insulin at baseline, oral antidiabetics (OAD), none).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Incretin Based Therapy (Randomized Group) | Insulin (Randomized Group) | Baseline Insulin (BL) (Non-randomized Group) | Oral Antidiabetic Drugs (OAD) (Non-randomized Group) | No OAD (Non-randomized Group)
Number analyzed (Participants) | 38 | 43 | 19 | 46 | 103
mg/dL
  Baseline: All Patients | 111.1 (18.95) | 111.8 (18.20) | 157.7 (66.50) | 97.2 (14.24) | 92.2 (8.58)
  Change at EOP: All Patients: number analyzed (Participants) | 37 | 41 | 19 | 45 | 101
  Change at EOP: All Patients | 22.2 (31.67) | 22.5 (34.05) | 9.8 (75.67) | 22.9 (23.40) | 16.3 (13.63)
  Baseline: Cushing's: number analyzed (Participants) | 12 | 13 | 6 | 13 | 15
  Baseline: Cushing's | 117.9 (20.99) | 106.3 (15.71) | 147.2 (68.38) | 93.3 (10.98) | 85.5 (6.92)
  Change at EOP: Cushing's: number analyzed (Participants) | 12 | 12 | 6 | 13 | 14
  Change at EOP: Cushing's | 13.4 (34.92) | 36.4 (33.11) | 21.3 (72.01) | 15.8 (18.43) | 11.7 (22.11)
  Baseline: Acromegaly: number analyzed (Participants) | 26 | 30 | 13 | 33 | 88
  Baseline: Acromegaly | 107.9 (17.46) | 114.2 (18.91) | 162.5 (67.85) | 98.8 (15.20) | 93.4 (8.32)
  Change at EOP: Acromegaly: number analyzed (Participants) | 25 | 29 | 13 | 32 | 87
  Change at EOP: Acromegaly | 26.5 (29.79) | 16.7 (33.29) | 4.6 (79.57) | 25.8 (24.82) | 17.0 (11.75)

7. Secondary Outcome: Percentage of Participants With ≤ 0.3% HbA1c Increase to End of Core Phase
Description: Percentage of participants with ≤ 0.3% HbA1c increase in the incretin based therapy arm and the insulin arm.
Time Frame: Randomization, up to 16 weeks
Population: Randomized Analysis Set (RAS): all participants who received at least one dose of pasireotide and were assigned to either incretin based therapy or insulin by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Incretin Based Therapy (Randomized Group) | Insulin (Randomized Group)
Number analyzed (Participants) | 38 | 43
Percentage of participants | 73.7 [56.9 to 86.6] | 65.1 [49.1 to 79.0]

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse Events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to approximately 46 months.
Description: There are different safety follow-up period for Cushing's and for acromegaly patients: On-treatment period: from day of first dose of study medication to 28 days after last dose of pasireotide s.c. and 84 days after last dose of pasireotide long acting, or the follow-up visit, whichever comes later.
Arm/Group | Incretin Based Therapy (Randomized Group) | Insulin (Randomized Group) | Baseline Insulin (BL) (Non-randomized Group) | Oral Antidiabetic Drugs (OAD) (Non-randomized Group) | No OAD (Non-randomized Group)
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/43 | 1/19 | 0/46 | 1/103
Serious Adverse Events (participants affected / at risk) | 6/38 | 3/43 | 4/19 | 2/46 | 7/103
Other Adverse Events (participants affected / at risk) | 37/38 | 40/43 | 18/19 | 38/46 | 87/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Incretin Based Therapy (Randomized Group) (N=38) | Insulin (Randomized Group) (N=43) | Baseline Insulin (BL) (Non-randomized Group) (N=19) | Oral Antidiabetic Drugs (OAD) (Non-randomized Group) (N=46) | No OAD (Non-randomized Group) (N=103)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Epiglottitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Tubular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 2
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Shock (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Incretin Based Therapy (Randomized Group) (N=38) | Insulin (Randomized Group) (N=43) | Baseline Insulin (BL) (Non-randomized Group) (N=19) | Oral Antidiabetic Drugs (OAD) (Non-randomized Group) (N=46) | No OAD (Non-randomized Group) (N=103)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 2 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 6
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 0 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 4 | 0 | 0 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 11 | 12 | 2 | 10 | 21
Erosive duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 13 | 7 | 0 | 5 | 11
Vomiting (Gastrointestinal disorders) | 5 | 0 | 0 | 2 | 1
Asthenia (General disorders) | 2 | 0 | 0 | 1 | 2
Fatigue (General disorders) | 4 | 4 | 0 | 1 | 5
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 5 | 8 | 0 | 4 | 9
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 1 | 3 | 1
Bone abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 4 | 0 | 3 | 16
Onychomycosis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 4
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 3 | 6 | 15
Urinary tract infection (Infections and infestations) | 3 | 5 | 1 | 0 | 4
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 2 | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 1 | 1 | 2
Bacterial test positive (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 1 | 1 | 5
Blood creatinine increased (Investigations) | 2 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 2 | 1 | 0 | 3 | 9
Blood insulin increased (Investigations) | 1 | 0 | 1 | 0 | 1
Blood urea increased (Investigations) | 1 | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 2 | 1 | 0 | 0
Carbon dioxide decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 4 | 0 | 2 | 0
Glycosylated haemoglobin increased (Investigations) | 3 | 1 | 0 | 0 | 1
Lipase increased (Investigations) | 3 | 2 | 0 | 1 | 5
Weight decreased (Investigations) | 10 | 4 | 0 | 5 | 2
Weight increased (Investigations) | 0 | 1 | 1 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 0 | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 9 | 2 | 14 | 4
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 14 | 11 | 6 | 9 | 13
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 10 | 8 | 5 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 2 | 0
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 14
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 2 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 4 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 5 | 5 | 0 | 3 | 6
Dysgeusia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 4 | 0 | 2 | 12
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 1 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT02060383/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT02060383/SAP_001.pdf